CLINICAL TRIAL: NCT03831347
Title: Adaptation and Pilot Study of Yoga to Reduce Depression in Adolescents
Brief Title: Treatments for Improving Mood in Depressed Teens-2
Acronym: TeenThrive
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brown University (Other)
Collaborators: Butler Hospital (Other); National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1801001977 Open; R34AT009886 (NIH)
Record Dates: First submitted 2019-01-30; First posted 2019-02-05 (Actual); Results first posted 2022-03-23 (Actual); Last update posted 2022-03-23 (Actual); Status verified 2022-02

CONDITIONS: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hatha Yoga (Experimental): 12 weeks of modified Hatha Yoga specifically designed to be administered to teens with depression.
  Interventions: Behavioral: Hatha Yoga

INTERVENTIONS:
Behavioral: Hatha Yoga — 12 weeks of Hatha Yoga

SUMMARY:
Phase 2: Open Trial N=12 adolescents will be enrolled into a single-arm pilot trial to test the adapted hatha yoga intervention

DETAILED DESCRIPTION:
In Phase 2, the investigators will conduct an open single-arm pilot trial of our 12 week adapted hatha yoga intervention.

the investigators will enroll 12 adolescents in the open pilot trial.

ELIGIBILITY:
Inclusion Criteria:

1. Adolescents must have elevated depressive symptoms, defined by a score of 11 or higher on the Quick Inventory of Depression -Adolescent Version-- Clinician Rating (QIDS-A-CR), including endorsement of either sad mood or anhedonia on the QIDS.
2. Other treatment for depression must be stable at baseline. Adolescents do not have to be in other treatment for depression, but, if they are, it must be stable for the past 12 weeks.
3. Adolescents must be aged 13-18.
4. Adolescents must be medically cleared for moderate physical activity by their primary care physician. This criterion may be met by a current (dated in the past year) statement from their pediatrician that the adolescent may participate in school or camp programs including physical education.
5. Adolescents must be able to read and write English sufficient to complete informed consent and engage in interventions.
6. Adolescents aged 13-17 must assent to be in the study, and their parent or legal guardian must consent to their participation. Adolescents aged 18 must consent to be in the study.
7. Able to attend one of the class times.

Exclusion Criteria:

1. QIDS- A-CR may not be higher than a score of 21. This ensures that adolescents are not severely depressed.
2. Adolescents who meet criteria for:

   * Current (past year) autism spectrum disorder (AS), if of sufficient severity to interfere with study treatment per clinician judgment;
   * Schizophrenia;
   * Bipolar disorder;
   * Clinically significant psychotic symptoms in the past month;
   * Anorexia or Bulimia in past 3 months
   * Substance use disorders in the past 12 months and symptoms are of sufficient severity to interfere with study treatment per clinician judgment These will be assessed with the Mini-International Neuropsychiatric Interview (MINI).
3. Adolescents may not have current suicide ideation or behavior that warrants immediate treatment. They may have passive ideation (i.e., thoughts that life is not worth living), but may not have active suicide ideation, intent, plan, or an attempt within the previous 6 months.
4. Adolescents cannot currently be engaged in or yoga classes, as this is the study intervention.
5. Adolescents cannot be pregnant as yoga should be modified for pregnancy

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 11 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2019-08-14 (Actual); Study Completion 2019-08-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Uebelacker, PhD, Principal Investigator — Butler Hospital; Shirley Yen, PhD, Principal Investigator — Brown University
Locations (1):
- Butler Hospital, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD underlying publication if required by journal.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: One year after study collection.
Access Criteria: Information available upon request, please send to PIs Lisa Uebelacker or Shirley Yen.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Hatha Yoga
Started | 11
Completed | 9
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | Hatha Yoga
Number analyzed (Participants) | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.8 (1.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 9
  Multiracial and Other | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 11

OUTCOME MEASURES:

1. Primary Outcome: Acceptability
Description: Acceptability assessed based on number of participants who remained in the intervention (retention).
Time Frame: Post intervention (month 3)
Population: Entire sample
Measure: Count of Participants; unit: Participants
Arm/Group | Hatha Yoga
Number analyzed (Participants) | 11
Participants | 9

2. Primary Outcome: Credibility Expectancy Questionnaire (CEQ) - Credibility Subscale
Description: Credibility assessed with Credibility Expectancy Questionnaire (CEQ), credibility subscale. The credibility subscale of the CEQ, is a 3 item subscale of the 6 item CEQ. The 3 items are scored on a range of 0-1. Higher scores indicate greater credibility.
Time Frame: Week 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Hatha Yoga
Number analyzed (Participants) | 11
score on a scale | 0.76 (0.25)

3. Primary Outcome: Credibility Expectancy Questionnaire (CEQ) - Expectancy Subscale
Description: Patient expectations assessed with the Credibility Expectancy Questionnaire (CEQ), expectancy subscale. The expectancy subscale is a 3 item subscale of the 6 item CEQ. Score ranges from 0-1 with higher scores indicating greater expectations.
Time Frame: Week 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Hatha Yoga
Number analyzed (Participants) | 11
score on a scale | 0.66 (0.29)

4. Primary Outcome: The Client Satisfaction Questionnaire (CSQ-8)
Description: Satisfaction with treatment assessed with The Client Satisfaction Questionnaire (CSQ-8). The CSQ-8 is an 8-item measure with each item measured on a 1-4 scale, and total score range from 8-32. Higher scores indicate greater client satisfaction.
Time Frame: Post intervention (month 3)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Hatha Yoga
Number analyzed (Participants) | 9
score on a scale | 26.2 (6.1)

5. Primary Outcome: Home Practice Questionnaire
Description: Number of participants who met criteria for home practice (target of two practices per week) as assessed with a home practice questionnaire.
Time Frame: Post intervention (month 3)
Measure: Count of Participants; unit: Participants
Arm/Group | Hatha Yoga
Number analyzed (Participants) | 10
Participants | 6

6. Primary Outcome: Systematic Assessment of Treatment-emergent Events-general Inquiry (SAFTEE)
Description: Participant safety/adverse events will be measured using the SAFTEE. Participants will also be asked weekly if they experienced any injuries as a result of yoga.
Time Frame: Post intervention (month 3)
Measure: Number; unit: adverse events
Arm/Group | Hatha Yoga
Number analyzed (Participants) | 11
adverse events | 6

7. Secondary Outcome: Quick Inventory of Depression - Adolescent Version - Clinician Rating (QIDS-A-CR)
Description: Depression symptom severity at Month 3. The QIDS is a 17 item measure with scores ranging from 0-30. Higher scores indicate greater depressive symptoms.
Time Frame: post intervention (month 3)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Hatha Yoga
Number analyzed (Participants) | 9
score on a scale | 4.11 (2.66)

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Hatha Yoga
All-Cause Mortality (participants affected / at risk) | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11
Other Adverse Events (participants affected / at risk) | 2/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hatha Yoga (N=11)
Infection (Blood and lymphatic system disorders) | 1 (2)
Celiac (Gastrointestinal disorders) | 1 (2)
GI distress (Gastrointestinal disorders) | 1 (1)
Gynecological issue (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-12-10): https://cdn.clinicaltrials.gov/large-docs/47/NCT03831347/Prot_SAP_000.pdf
  • Informed Consent Form (2019-04-17): https://cdn.clinicaltrials.gov/large-docs/47/NCT03831347/ICF_001.pdf